CLINICAL TRIAL: NCT07155226
Title: A Modular Phase I/II, Open-label, Multi-Centre Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of AZD3632 Monotherapy or in Combination With Anticancer Agents in Participants With Advanced Haematologic Malignancies With KMT2Ar, NPM1m, or Other Genotypes Associated With HOX Overexpression
Brief Title: Study of AZD3632 Monotherapy or in Combination With Anticancer Agents in Participants With Advanced Haematologic Malignancies With KMT2Ar, NPM1m, or Other Genotypes Associated With HOX Overexpression
Acronym: MOMENTUM
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D8620C00001; 2025-521299-76-00 (Other: EU CT number)
Record Dates: First submitted 2025-08-14; First posted 2025-09-04 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Acute Lymphoblastic Leukaemia; Acute Myeloid Leukaemia; Higher-risk Myelodysplastic Syndromes
Keywords: Myelodysplastic Syndromes; Menin inhibitor; Anti-leukaemic activity; Anti-fungal agent; HOX overexpression.
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — posaconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Module 1: AZD3632 dose 1 (Experimental): Participants will receive AZD3632 (dose 1) through the treatment period.
  Interventions: Drug: AZD3632
- Module 1: AZD3632 dose 2 (Experimental): Participants will receive AZD3632 (dose 2) through the treatment period.
  Interventions: Drug: AZD3632
- Module 1: AZD3632 dose 3 (Experimental): Participants will receive AZD3632 (dose 3) through the treatment period.
  Interventions: Drug: AZD3632
- Module 1: AZD3632 dose 4 (Experimental): Participants will receive AZD3632 (dose 4) through the treatment period.
  Interventions: Drug: AZD3632
- Module 1: AZD3632 dose 5 (Experimental): Participants will receive AZD3632 (dose 5) through the treatment period.
  Interventions: Drug: AZD3632
- Module 1: AZD3632 dose 6 (Experimental): Participants will receive AZD3632 (dose 6) through the treatment period.
  Interventions: Drug: AZD3632
- Module 2: AZD3632 + posaconazole (Experimental): Participants will receive AZD3632 alone, then will receive AZD3632 in combination with posaconazole through treatment period.
  Interventions: Drug: AZD3632; Drug: Posaconazole

INTERVENTIONS:
Drug: AZD3632 — AZD3632 will be administered orally.
Drug: Posaconazole — Posaconazole will be administered orally.
  Arms: Module 2: AZD3632 + posaconazole

SUMMARY:
The purpose of this study is to understand the safety, tolerability, efficacy, pharmacokinetic (PK), pharmacodynamic (PD), and preliminary efficacy of orally administered AZD3632 in participants with advanced haematologic malignancies with KMT2Ar, NPM1m, or other genotypes associated with homeobox (HOX) overexpression.

DETAILED DESCRIPTION:
This is a first in human (FTiH), open-label, multi-centre study of AZD3632 in participants with relapsed or refractory acute leukaemia or myelodysplastic Syndromes (MDS) with HOX overexpression genotypes.

This study includes multiple modules (module 1 and module 2) each investigating AZD3632 in a specific population and/or in combination with other anticancer agents.

Module 1 is a dose escalation of AZD3632 monotherapy. Module 2 will investigate the safety, PK, and tolerability when co-administered with posaconazole.

ELIGIBILITY:
Key Inclusion Criteria:

Core criteria:

* Adequate organ function.
* Contraceptive use by participants or participant partners should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Module 1:

* Advanced haematologic malignancy - a) for dose escalation - diagnosis of acute leukemia or myelodysplastic neoplasia (MDS) and harbouring one of the genetic alterations per local testing associated with upregulation of HOX; b) for Backfill - diagnosis of harbouring a KMT2Ar or NPM1m per local testing.
* Participants must have measurable disease that is relapsed/refractory to conventional therapies known to be effective for their disease and not have any available approved therapies.: a) Relapsed and primary refractory acute leukaemia after standard of care therapy including but not limited to 2 cycles of intensive chemotherapy, hypomethylating agent (HMA) monotherapy, or HMA combinations such as HMA/venetoclax.; b) Relapsed and primary refractory MDS is defined by ≥ 5% blasts in the bone marrow and/or persistence of peripheral blasts after treatment with at least 2 cycles of HMA. Participants ineligible for the treatment with an HMA and without any other standard of care (SoC) options are allowed to enrol; c) White blood cell count below 25,000/μL. Participants may receive cytoreduction per protocol-specified criteria; d) Performance status: Eastern Cooperative Operative Group (ECOG) ≤ 2; e) Life expectancy: ≥ 8 weeks.

Module 2:

* Participants must have measurable disease that is relapsed/refractory to conventional therapies known to be effective for their disease and not have any available approved therapies.: a) Relapsed and primary refractory acute leukaemia after standard of care therapy including but not limited to 2 cycles of intensive chemotherapy, HMA monotherapy, or HMA combinations such as HMA/venetoclax.; b) Relapsed and primary refractory MDS is defined by ≥ 5% blasts in the bone marrow and/or persistence of peripheral blasts after treatment with at least 2 cycles of HMA. Participants ineligible for the treatment with an HMA and without any other SoC options are allowed to enrol; c) White blood cell count below 25,000/μL. Participants may receive cytoreduction per protocol-specified criteria; d) Performance status: ECOG ≤ 2; e) Life expectancy: ≥ 8 weeks.

Key Exclusion Criteria:

Core criteria:

* Participants with Burkitt lymphoma/leukaemia or Acute Promyelocytic Leukaemia.
* Active testicular or active central nervous system (CNS) (> CNS1 or radiographic) involvement by leukaemia.
* Unresolved treatment-related toxicities Grade ≥ 2 from prior therapy.
* Abnormal levels of potassium or magnesium prior to first dose of AZD3632.

Module 1:

* Receipt of non-CNS radiation therapy within 2 weeks and of CNS radiation within 8 weeks of the first scheduled dose.
* Receipt of any investigational or non-investigational anticancer agents, including non-biologic agents, biologic agents and/or prior treatment other menin inhibitors (backfill participants only).
* For nested food effect participants - diagnosis of diabetes mellitus (Type I or Type II).

Module 2:

* Receipt of any non-investigational anticancer agents, including non-biologic agents and/or biologic agents or receipt of non-CNS or CNS radiation therapy.
* Participants for whom treatment with posaconazole is contraindicated per the local prescribing information.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2026-01-09 (Actual); Primary Completion 2029-02-15 (Estimated); Study Completion 2029-02-15 (Estimated)

PRIMARY OUTCOMES:
Module 1: Number of participants with dose-limiting toxicity (DLT) | At the end of Cycle 1 (each cycle is 28 days)
  Safety and tolerability of AZD3632 monotherapy in participants with advanced haematologic malignancies will be assessed.
Module 1 and Module 2: Number of participants with dose modification, delay and discontinuations due to adverse events (AEs) | Up to 3 years 1 month
  Safety and tolerability of AZD3632 monotherapy in participants with advanced haematologic malignancies will be assessed.
Module 1 and Module 2: Number of participants with treatment-emergent adverse events (TEAEs), treatment-related AEs (TRAEs) and serious adverse vents (SAEs) | Up to 30 days after last dose (approximately 3 years 1 month)
  Safety and tolerability of AZD3632 monotherapy in participants with advanced haematologic malignancies will be assessed. Adverse events will be defined as treatment-emergent if they have an onset or worsen (by investigator report of a change in intensity) during the study treatment or the safety follow-up period but prior to any subsequent cancer therapy.

SECONDARY OUTCOMES:
Module 1 and Module 2: Maximum concentration (Cmax) of AZD3632 | From Day 1 to 3 years 1 month
  The PK of AZD3632 as monotherapy (module 1) and in combination with posaconazole (module 2) will be assessed.
Module 1 and Module 2: Time of maximum concentration (Tmax) of AZD3632 | From Day 1 to 3 years 1 month
  The PK of AZD3632 as monotherapy (module 1) and in combination with posaconazole (module 2) will be assessed.
Module 1: Trough concentration (Ctrough) of AZD3632 | From Day 1 to 3 years 1 month
  The PK of AZD3632 as monotherapy will be assessed.
Module 1: Area under the plasma concentration-time Curve from Time Zero to Infinity (AUC[inf]) of AZD3632 | From Day 1 to 3 years 1 month
  The PK of AZD3632 as monotherapy will be assessed.
Module 1 and Module 2: Area under the curve from time 0 to the time of last measurable concentration (AUC[0-t]) of AZD3632 | From Day 1 to 3 years 1 month
  The PK of AZD3632 as monotherapy (module 1) and in combination with posaconazole (module 2) will be assessed.
Module 1: Area under concentration-time curve in the dosing interval (AUCtau) of AZD3632 | From Day 1 to 3 years 1 month
  The PK of AZD3632 as monotherapy will be assessed.
Module 1: Apparent total body clearance (CL/F) of AZD3632 | From Day 1 to 3 years 1 month
  The PK of AZD3632 as monotherapy will be assessed.
Module 1: Apparent volume of distribution based on the terminal phase (VZ/F) of AZD3632 | From Day 1 to 3 years 1 month
  The PK of AZD3632 as monotherapy will be assessed.
Module 1: Half-life (t1/2) of AZD3632 | From Day 1 to 3 years 1 month
  The PK of AZD3632 as monotherapy will be assessed.
Module 1: Maximum concentration (Cmax) of AZD3632 (food effect) | From Day 1 to 3 years 1 month
  The preliminary effect of food on plasma PK of AZD3632 (conducted in a nested evaluation during backfills) will be assessed.
Module 1: Time of maximum concentration (Tmax) of AZD3632 (food effect) | From Day 1 to 3 years 1 month
  The preliminary effect of food on plasma PK of AZD3632 (conducted in a nested evaluation during backfills) will be assessed.
Module 1 and Module 2: Area under the curve from time 0 to the time of last measurable concentration (AUC[0-t]) of AZD3632 (food effect) | From Day 1 to 3 years 1 month
  The preliminary effect of food on plasma PK of AZD3632 (conducted in a nested evaluation during backfills) will be assessed.
Module 1: Area under concentration-time curve in the dosing interval (AUCtau) of AZD3632 (food effect) | From Day 1 to 3 years 1 month
  The preliminary effect of food on plasma PK of AZD3632 (conducted in a nested evaluation during backfills) will be assessed.
Module 1: Minimum concentration (Cmin) of AZD3632 (food effect) | From Day 1 to 3 years 1 month
  The preliminary effect of food on plasma PK of AZD3632 (conducted in a nested evaluation during backfills) will be assessed.
Module 1: Ratio of Cmax between fed and fasted state | From Day 1 to 3 years 1 month
  The preliminary effect of food on plasma PK of AZD3632 (conducted in a nested evaluation during backfills) will be assessed.
Module 1: Ratio of AUC(0-t) between fed and fasted state | From Day 1 to 3 years 1 month
  The preliminary effect of food on plasma PK of AZD3632 (conducted in a nested evaluation during backfills) will be assessed.
Module 1: Ratio of AUCtau between fed and fasted state | From Day 1 to 3 years 1 month
  The preliminary effect of food on plasma PK of AZD3632 (conducted in a nested evaluation during backfills) will be assessed.
Module 2: Plasma geometric mean ratio of Cmax | From Day 1 to 3 years 1 month
  The PK pf AZD3632 when co-administered with posaconazole will be assessed.
Module 2: Plasma geometric mean ratio of AUC | From Day 1 to 3 years 1 month
  The PK pf AZD3632 when co-administered with posaconazole will be assessed.
Module 2: Plasma concentration of posaconazole | From Day 1 to 3 years 1 month
  The PK pf AZD3632 when co-administered with posaconazole will be assessed.
Module 1 and Module 2: Complete response rate (CR + CRh) | Up to 3 years 1 month
  Complete response rate is defined as the percentage of participants who have a complete remission (CR) or complete remission with partial haematological recovery (CRh) as assessed by the investigator at local site.
Module 1 and Module 2: Time to response (TTR) | Up to 3 years 1 month
  TTR in participants with acute leukaemia is defined as the time from date of first dose until date of first documented complete response (CR/CRh) among participants with acute leukaemia in the Response Evaluable Set who achieved complete response as assessed by investigator at local site.
  TTR in participants with MDS is defined as the time from date of first dose until date of first documented objective response a CR (or CR equivalent), complete response with limited count recovery [CRL], CRh, partial response [PR], or haematologic improvement [HI]) among participants with MDS in the Response Evaluable Set who achieved objective response as assessed by investigator at local site.
Module 1 and Module 2: Duration of response (DoR) | Up to 3 years 1 month
  DoR in participants with acute leukaemia is defined as the time from date of first documented complete response (CR/CRh) until date of first documented relapse or death (by any cause in the absence of relapse) as assessed by investigator at local site.
  DoR in participants with MDS is defined as the time from date of first documented objective response CR (or CR equivalent), CRL, CRh, PR, or HI until date of first documented relapse or death (by any cause in the absence of relapse) as assessed by investigator at local site.
Module 1 and Module 2: Transfusion Independence (TI) | Up to 3 years 1 month
  TI is defined as no RBC and no platelet transfusion during any consecutive period of at least 56 days post-baseline after starting treatment with AZD3632 or cessation of treatment with AZD3632 but prior to start of subsequent new therapy.
Module 1 and Module 2: Event-free Survival (EFS) | From Cycle 2 Day 1 (each cycle is 28 days) up to disease follow-up (approximately 3 years 1 month)
  EFS for participants with acute leukaemia is defined as the time from date of first dose until date of relapse, progressive disease, failure to achieve at least Morphologic leukaemia-free state (MLFS) by end of Cycle 6, or death due to any cause as assessed by investigator at a local site.
  EFS for participants with MDS is defined as the time from date of first dose until date of relapse, progressive disease, failure to achieve at least HI by end of Cycle 6, or death due to any cause.
Module 1 and Module 2: Overall Survival (OS) | From Cycle 2 Day 1 (each cycle is 28 days) up to disease follow-up (approximately 3 years 1 month)
  OS is defined as the time from date of first dose until date of death due to any cause regardless of whether the participant withdraws from study therapy or receives another anticancer therapy.
Module 1 and Module 2: Percentage of participants who receive subsequent allogeneic hematopoietic stem cell transplant (HSCT) | Up to 3 years 1 month
  Percentage of participants with acute leukaemia and MDS who receive subsequent allogeneic HSCT will be reported.
Module 1 and Module 2: Overall Response Rate (ORR) | Up to 3 years 1 month
  ORR in participants with myelodysplastic syndromes (MDS) is defined as the percentage of participants who have a CR (or CR equivalent), CRL, CRh, PR, or HI as determined by investigator at a local site.
Module 1 and Module 2: Time to Progression to acute myeloid leukaemia (AML) | Up to 3 years 1 month
  Time to progression to AML is defined from the time of first dose of AZD3632 until first diagnosis of AML, regardless of discontinuation of treatment or receiving of subsequent therapy.

CONTACTS AND LOCATIONS:
Locations (26):
- United States (5):
  - Research Site, Decatur, Illinois
  - Research Site, New York, New York
  - Research Site, Durham, North Carolina
  - Research Site, Portland, Oregon
  - Research Site, Houston, Texas
- Australia (2):
  - Research Site, Fitzroy
  - Research Site, Perth
- Canada (2):
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- Research Site, Copenhagen, Denmark
- Germany (6):
  - Research Site, Dresden
  - Research Site, Frankfurt A. Main
  - Research Site, Halle
  - Research Site, Heidelberg
  - Research Site, München
  - Research Site, Ulm
- Italy (2):
  - Research Site, Bologna
  - Research Site, Ravenna
- Japan (3):
  - Research Site, Bunkyō City
  - Research Site, Kashiwa
  - Research Site, Okayama
- Research Site, Seoul, South Korea
- United Kingdom (4):
  - Research Site, Edinburgh
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Newcastle

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portalVivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure."Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitment a made to the EFPIA PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/